CLINICAL TRIAL: NCT02056743
Title: Clinical Trials on Evaluate the Red Ginseng and Fermented-Red Ginseng Affect to Drug Metabolizing Enzyme and Transporter in Healthy Volunteers; Open-label, Parallel Group
Brief Title: Clinical Trials on Evaluate the Red Ginseng and Fermented-Red Ginseng Affect to Drug Metabolizing Enzyme and Transporter in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Dal-Sik Kim, Professor, MD, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CUH_2012_RG
Record Dates: First submitted 2014-02-02; First posted 2014-02-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
MeSH Terms: interventions — Caffeine; Losartan; Omeprazole; Dextromethorphan; Midazolam; fexofenadine; Asian ginseng

ARMS (2):
- Fermented-red ginseng (Experimental): At period 1, the fermented-red ginseng group administered CYP cocktail (Caffeine 200mg + Losartan 50mg + Omeprazole 20mg + Dextromethorphan 30mg + Midazolam 7.5mg) under fasting conditions on the first day. At second day, they administered Fexofenadine 30mg under fasting conditions.
  During 4~17th days they administered fermented-red ginseng. At period 2, the fermented-red ginseng group administered CYP cocktail (Caffeine 200mg + Losartan 50mg + Omeprazole 20mg + Dextromethorphan 30mg + Midazolam 7.5mg) under fasting conditions on the 15th day. At 16th day, they administered Fexofenadine 30mg under fasting conditions.
  Interventions: Drug: CYP cocktail; Drug: Fexofenadine 30mg; Dietary Supplement: Fermented-red ginseng
- Red ginseng (Experimental): At period 1, the red ginseng group administered CYP cocktail (Caffeine 200mg + Losartan 50mg + Omeprazole 20mg + Dextromethorphan 30mg + Midazolam 7.5mg) under fasting conditions on the first day. At second day, they administered Fexofenadine 30mg under fasting conditions.
  During 4~17th days they administered red ginseng. At period 2, the red ginseng group administered CYP cocktail (Caffeine 200mg + Losartan 50mg + Omeprazole 20mg + Dextromethorphan 30mg + Midazolam 7.5mg) under fasting conditions on the 15th day. At 16th day, they administered Fexofenadine 30mg under fasting conditions.
  Interventions: Drug: CYP cocktail; Drug: Fexofenadine 30mg; Dietary Supplement: Red ginseng

INTERVENTIONS:
Drug: CYP cocktail — Each group administered CYP cocktail (Caffeine 200mg + Losartan 50mg + Omeprazole 20mg + Dextromethorphan 30mg + Midazolam 7.5mg) under fasting conditions.
  Other Names: Caffeine 200mg; Losartan 50mg; Omeprazole 20mg; Dextromethorphan 30mg; Midazolam 7.5mg
Drug: Fexofenadine 30mg — Each group administered Fexofenadine 30mg under fasting conditions.
Dietary Supplement: Red ginseng — During 4~17th days, end of the period 1, the group of red ginseng administered red ginseng extract.
  Arms: Red ginseng
Dietary Supplement: Fermented-red ginseng — During 4~17th days, end of the period 1, the group of fermented-red ginseng administered fermented-red ginseng extract.
  Arms: Fermented-red ginseng

SUMMARY:
The purpose of this study is to evaluate the possibility of drug interactions before and after taking red ginseng or fermented-red ginseng by estimating metabolic rate of indicator drugs for cytochrome P450 and P-glycoprotein.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 20 and 55 years.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight > 45 kg.
* An informed consent document signed and dated by the subject.
* Subject who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
* Any condition possibly affecting drug absorption (e.g. gastrectomy)
* History of regular alcohol consumption exceeding 21 drinks/week (1 drink = 150 mL of wine or 360 mL of beer or 45 mL of hard liquor) within 6 months of Screening
* Participating in a bioequivalence study or other clinical study within 3 months preceding the first dose of study medication
* Screening sitting blood pressure > 160 mm Hg (systolic) or >90 mm Hg (diastolic), following at least 5 minutes of rest.
* History of significant alcohol abuse or drug abuse within one year prior to the Screening
* Use of any drugs known to significantly induce or inhibit drug-metabolizing enzymes within 30 days prior to dosing
* Smoking over 20 cigarettes per day
* Use of prescription or nonprescription drugs and dietary supplements within 10 days or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* Blood donation within 2 months prior to dosing, or plasma donation within 2 weeks prior to dosing
* Unwilling or unable to comply with the Lifestyle guidelines described in this protocol
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study
* Subjects who are hypersensitive to investigational drugs or related compounds
* Subjects with hereditary disease of galactose intolerance, Lapp lactase deficiency or gulucose-galactose malabsorption
* Subjects who are decided incongruity to participated in this study by investigators

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | CYP cocktail: 0, 0.25, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 h / Fexofenadine: 0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 h
Area under the plasma concentration curve (AUClast) | CYP cocktail: 0, 0.25, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 h / Fexofenadine: 0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 h

SECONDARY OUTCOMES:
Area under the plasma concentration curve (AUCinf) | CYP cocktail: 0, 0.25, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 h / Fexofenadine: 0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 h
First time to reach Cmax (Tmax) | CYP cocktail: 0, 0.25, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 h / Fexofenadine: 0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 h
Terminal half-life (t1/2) | CYP cocktail: 0, 0.25, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 h / Fexofenadine: 0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 h
Apparent Total Body Clearance (CL/F) | CYP cocktail: 0, 0.25, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 h / Fexofenadine: 0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 h
Apparent Volume of Distribution (Vd/F) | CYP cocktail: 0, 0.25, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 h / Fexofenadine: 0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 h

OTHER OUTCOMES:
AUClast ratio | Up to last analysis time of each drug and concentration ratio of drug/metabolite in plasma and urine samples of various sampling time
  CYP cocktail: 0, 0.25, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 h / Fexofenadine: 0, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 h / Urine for Losartan and Dextromethorphan: 0-4, 4-8, 8-12 h

CONTACTS AND LOCATIONS:
Overall Officials: Dal-Sik Kim, PhD, MD, Principal Investigator — Laboratory medicine; Min-Gul Kim, MD, Principal Investigator — Biomedical Research Institute
Locations (1):
- Clinical Trial Center of Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

REFERENCES:
- [Derived] Kim DS, Kim Y, Jeon JY, Kim MG. Effect of Red Ginseng on cytochrome P450 and P-glycoprotein activities in healthy volunteers. J Ginseng Res. 2016 Oct;40(4):375-381. doi: 10.1016/j.jgr.2015.11.005. Epub 2015 Dec 17. PMID 27746690
- [Derived] Kim MG, Kim Y, Jeon JY, Kim DS. Effect of fermented red ginseng on cytochrome P450 and P-glycoprotein activity in healthy subjects, as evaluated using the cocktail approach. Br J Clin Pharmacol. 2016 Dec;82(6):1580-1590. doi: 10.1111/bcp.13080. Epub 2016 Oct 9. PMID 27495955